CLINICAL TRIAL: NCT03211624
Title: The Etiology and Extent of Impaired Quality of Life, Fatigue and Cognitive, Affective and Emotional Dysfunction in Patients With Cushing's Syndrome - Prospective Studies
Brief Title: Quality of Life, Fatigue and Cognitive, Affective and Emotional Dysfunction in Patients With Cushing's Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Leiden University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: CognCush
Record Dates: First submitted 2017-06-14; First posted 2017-07-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Cushing Syndrome
MeSH Terms: conditions — Cushing Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples for DNA and RNA isolation will be collected and stored at -80°C.
  Polymorphism in the glucocorticoid (GC) receptor gene, and other genes involved in metabolism and transport of GCs will be analysed in all subjects at inclusion in the study.
  DNA methylation and mRNA will be analyzed at inclusion and 24 months after treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cushing syndrome: Male and female patients with Cushing syndrome caused by ACTH-producing pituitary adenoma or cortisol producing adrenal adenoma
- Controls: Healthy controls matched for age, gender, and educational level

SUMMARY:
This is a prospective, multi-center, case-control study where neurocognitive function will be evaluated in 36 patients with Cushing syndrome (CS) and 36 controls matched for age, gender and education.

DETAILED DESCRIPTION:
1. Background

   Endogenous Cushing's syndrome (CS) is the collective name for several rare disorders of chronic glucocorticoid (GC) excess. The most common causes are ACTH producing pituitary adenoma [Cushing's disease (CD)], cortisol producing adrenal adenoma (CPAA) and ectopic ACTH producing tumors.

   Cognitive dysfunction, psychiatric disorders, fatigue, and impaired quality of life (QoL) are frequently observed in patients with active CS. Morphological changes in the central nervous system have also been reported in patients with CS, including decreased total brain volume and hippocampal formation volume compared with healthy subjects.

   After successful treatment of CS, cognitive function improves according to some studies while others have found no change from pre-treatment levels. Increased brain volume has also been reported following treatment, although not to the levels of a normal control group.

   Various aspects of the neurocognitive consequences of hypercortisolism have been studied in recent years. However, a major limitation of most previous studies is the small sample size. Longitudinal research data is sparse. A further limitation is that CS is a heterogeneous disease with several etiologies, varied clinical findings at presentation and varying outcome after treatment. Consequently, and since CS is a rare syndrome, the number of patients needed to be studied is too large for a single center. A collaborative multi-centre effort is therefore a desirable approach.
2. Aim

   The overall aims of this project are 1) to improve our understanding of CS, in particular the spectra and time course of impaired well-being, fatigue and cognition, 2) to study the mechanisms behind the apparently long-term negative consequences on the CNS in these domains after biochemical remission has been achieved. For this purpose, the investigators will use the following tools:
   * Structural MRI. To evaluate total brain volume and volume of structures important for cognitive function such as hippocampus and frontal cortex.
   * Diffusion Tensor Imaging (DTI). To evaluate structural connectivity and integrity of white matter
   * Resting state and task related functional MRI (fMRI). To evaluate brain functional connectivity during rest and during testing of cognitive and emotional functioning. Primary regions of interests are the hippocampus, the frontal cortex and other key regions of the limbic circuitry.
   * Fludeoxyglucose Positron emission tomography (FDG-PET). To study glucose utilization in the above mentioned brain regions.
   * CSF analysis. To understand the significance of inflammatory and neurodegenerative biomarkers in CSF and blood in patients with CS.
   * Genetic and epigenetic analysis. To evaluate the influence of polymorphisms in the GC receptor gene, and genes involved in metabolism and transport of GCs, on cognitive and emotional functioning in patients with CS.
3. Design

   This is a prospective, case-controlled study, conducted at three centres:
   * The Department of Endocrinology, Sahlgrenska University Hospital, Gothenburg, Sweden.
   * The Department of Endocrinology/Medicine, Hospital Sant Pau, Barcelona, Spain.
   * The Department of Medicine, Division of Endocrinology, and Leiden Institute for Brain and Cognition/Department of Psychiatry, Leiden University Medical Center, Leiden, The Netherlands.

   Patients and matched controls will be recruited at each centre.

   The patients will be studied prior to medical and surgical treatment (baseline visit 0) and 3, 6, 9, 12, 18 and 24 months after surgical treatment. The controls will be studied on two occasions, namely at baseline and after 12 months.
4. Subjects Thirty-six patients with newly diagnosed endogenous CS and 36 matched controls will participate in the study.

   Since CS is a rare disorder the investigators estimate that it will take 3 years to include 36 patients.
5. Methods

   5.1 Inclusion

   The study investigators at each individual centre will identify patients with newly diagnosed CS. Inclusion will take place before any intervention, including medical treatment for hypercortisolism.

   5.2 Questionnaires

   Questionnaires will be completed by patients at the individual centres in the morning 9-12 am, prior to treatment and 6, 12 and 24 months after treatment. Controls will complete the questionnaires at baseline and after 12 months.
   1. The fatigue impact scale (FIS) will be used to evaluate fatigue.
   2. The EuroQol and CushingQoL will be used to evaluate quality of life.
   3. The Beck Depression Inventory and Beck Anxiety Inventory will be used to evaluate depression and anxiety
   4. The apathy scale will be used to evaluate apathy.

   5.3 Cognitive function

   The Rey Complex Figure will be used to test memory. Digit symbol-coding from the WAIS-IV NI will be used to assess information processing speed. Auditory attention and working memory will be measured by the digit span test. The verbal fluency test (FAS) will be used to measure the ability to generate as many words as possible beginning with a specific letter within 1 minute.

   5.4 Structural MRI (Magnetic Resonance Imaging)

   Patients will undergo cranial magnetic resonance imaging before treatment as well as 12 and 24 months after surgery. Control subjects will be scanned twice with an interval of approximately 12 months. In line with previous MRI studies in patient populations, total time for participants in the scanner will be one hour or less.

   5.5 Diffusion Tensor Imaging (DTI)

   The investigators will also acquire DTI data along 32 directions, enabling analyses of integrity as well as fibre tracking.

   5.6 Functional MRI

   Functional MRI will be used to study resting state functional connectivity as well as brain activity during cognitive and emotional function prior to treatment, and 12 and 24 months after treatment.

   5.7 Positron emission tomography

   Resting state glucose utilization in the brain will be studied by using fludeoxyglucose positron emission tomography (FDG-PET) prior to treatment and 12 months after treatment (only in patients from Gothenburg). Controls will be studied with FDG-PET only at baseline.

   5.8 Neurodegenerative and inflammatory biomarkers in CSF and blood

   Neurodegenerative and neuroinflammatory CSF markers, as well as peptides and hormones important for GC metabolism, will be analysed prior to treatment and 12 months after treatment (only in Gothenburg). Controls will be studied only at baseline.

   5.9 Genetics

   Polymorphism in the GC receptor gene, and other genes involved in metabolism and transport of GCs will be analysed in all subjects at inclusion in the study. All genetic analysis will be performed at Sahlgrenska University Hospital, Gothenburg, Sweden, in a single run at the end of the study.

   Blood samples for DNA and RNA will be collected at baseline and 24 months after treatment for analysis of methylation and mRNA expression.
6. Ethical considerations

   The study will be conducted according to the Declaration of Helsinki. Application for Ethical approval will be applied from the local ethical committees in Barcelona, Gothenburg and Leiden. Informed written consent will be obtained from all patients and controls. Incidental findings of clinical significance will be investigated further by the respective participating centers.
7. Statistical methods - Power calculations A power analysis based on previous results from studies on cognitive function as well as fMRI findings in patients with Cushing syndrome suggests that between 14 and 28 subjects need to be included in the study to detect a difference between patients with CS in remission and controls with a significance level of 5% and power of 80%. Because multiple comparisons will be applied, comparing brain activity between different groups on three performance tasks as well as a resting state condition, 36 participants per group will be included.
8. Financial disclosure

An unrestricted grant has been provided by HRA Pharma.

ELIGIBILITY:
Inclusion criteria:

* Male and female patients with Cushing syndrome (CS) caused by ACTH-producing pituitary adenoma or cortisol producing adrenal adenoma
* Age between 18 and 65 years

Exclusion criteria

* CS caused by ectopic ACTH producing tumours
* CS caused by adrenocortical carcinoma
* Pseudo CS
* Subclinical CS
* Exogenous CS
* Previous history of major psychiatric disorder (not related to CS)
* Neurological disorders affecting the central nervous system
* High alcohol consumption (more than 14 units of alcohol per week)
* Active malignancy or any treatment for malignancy during the last 2 years
* Heart failure (NYHC II-IV)
* Severe respiratory insufficiency
* Severely impaired hepatic function (alanine transaminase and/or aspartate transaminase concentrations two times the upper limit of normal or above)
* Severely impaired renal function (serum- creatinine >150 µmol/L or glomerular filtration rate <45 ml/min)
* Pregnancy or breast feeding
* Any other illness that significantly affects the patients cognitive function according to the investigators opinion
* Contraindication for MRI (Presence of medical implants, metal in the body, claustrophobia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty-six patients with newly diagnosed endogenous Cushing syndrome and 36 matched controls
Sampling Method: Probability Sample
Enrollment: 72 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Cognitive function | 2 years
  Improvement in memory 2 years after treatment of Cushing syndrome evaluated with the Rey Complex Figure.

SECONDARY OUTCOMES:
Test score in CushingQoL test | 2 years
  Improvement in quality of life 2 years after treatment of Cushing syndrome, measured with the CushingQoL, where total score at baseline and at 2 years will be compared by using the Wilcoxon signed-rank test.
Brain volume | 2 years
  Changes in total brain volume and volume of structures important for cognitive function such as hippocampus and frontal cortex 2 years after treatment of Cushing syndrome by using structural MRI
Functional brain response | 2 years
  Changes in brain functional connectivity during rest and during testing of cognitive and emotional functioning 2 years after treatment of Cushing syndrome by using functional MRI
Glucose utilization | 2 years
  Change in glucose utilization in the hippocampus and frontal cortex 2 years after treatment of Cushing syndrome by using Fludeoxyglucose Positron emission tomography (FDG-PET).
Polymorphisms in the GC receptor gene or genes involved in metabolism and transport of GCs | 2 years
  To evaluate the influence of polymorphisms in the GC receptor gene, and genes involved in metabolism and transport of GCs, on memory and attention in patients with CS.

CONTACTS AND LOCATIONS:
Overall Officials: Oskar Ragnarsson, MD, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (3):
- Dept of Medicine, Division of Endocrinology, and Center for Endocrine Tumors, Leiden University Medical Center, Leiden, Netherlands
- Dept of Endocrinology, Hospital Sant Pau, Barcelona, Spain
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
All data will be available for other researcher upon request.